CLINICAL TRIAL: NCT05412706
Title: Niraparib Maintenance Treatment in Metastatic Colorectal Cancer Patients With a Partial or Complete Response After Oxaliplatin-based Induction Therapy: Bohème Trial
Brief Title: Niraparib Maintenance Treatment in mCRC With a Partial o Complete Response After Oxaliplatin-based Induction Therapy
Acronym: Bohème
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The Principal Investigator has retired and has not been replaced has retired and a new one has not been identified Principal Investigator
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: CRO "Centro Clinical Trials" IRCCS Ospedale Policlinico San Martino (Unknown); Laboratory Molecular Oncology Candiolo Cancer Institute IRCCS - Candiolo (Torino) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bohème
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Niraparib metastatic colorectal cancer PARP1 PARP2 inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Treatment with Niraparib must be started after at least 2 weeks and no later than 6 weeks after the end of platinum-based induction therapy.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Patients will receive Niraparib 200-300 mg orally as an individualized weight and platelet-based, flat-fixed, continuous daily dose.
  Niraparib will be administered orally once daily in 28-day cycles.
  Other Names: Zejula

SUMMARY:
Colorectal Cancer ranks third among the most frequent malignancies representing a leading cause of cancer-related death worldwide. The constant improvement in the "continuum of care" of metastatic colorectal cancer (mCRC) patients led to a median overall survival of about 30-36 months.

Due to the cumulative toxicities of first-line combinations of chemotherapy and biological agents, discontinuation or intermittent chemotherapy or maintenance strategies have been investigated in clinical trials. After a 4 to 6-month induction treatment with bevacizumab plus doublet or triplet regimens, a fluoropyrimidine plus bevacizumab is regarded as the optimal maintenance regimen. Little evidence is available on the role of maintenance with anti-EGFR agents.

A recent systematic review and network meta-analysis of 12 relevant randomized clinical trials comprising 5540 patients with mCRC showed that a maintenance strategy with a fluoropyrimidine, with or without the addition of bevacizumab, is preferred. However, given the lack of a clear overall survival benefit, shared decision-making should include observation as an acceptable alternative.

Poly(ADP)-ribose polymerase (PARP) inhibitors are now approved for breast, ovarian and pancreatic cancers. Evidence suggests that PARP inhibitors are more effective in tumors harboring homologous recombination DNA damage repair (HRR) deficiency and platinum sensitivity may be used a surrogate marker of HRD and therefore of PARP-inhibitors efficacy. An extensive Next Generation Sequencing analysis revealed that 15% of mCRC samples harbors mutations in genes involved in the HRR pathway. Several clinical trials are ongoing to test PARP inhibitors either alone or in combination in mCRC patients. The originality of this trial is to investigate PARPi in the maintenance setting.

Pre-clinical evidence showed that PARP blockade after initial oxaliplatin response delayed disease progression in mCRC carrying Kirsten Rat Sarcoma and BRAF mutations, suggesting that maintenance treatment with PARP inhibitors warrants further clinical investigation in mCRC patients who respond to oxaliplatin-containing induction treatment.

The main objective of this trial is to investigate the efficacy of anti-PARP inhibition as maintenance treatment in mCRC patients who obtained a complete or partial response after 4-month induction treatment with oxaliplatin-based double or triplet plus biologic agents.

DETAILED DESCRIPTION:
Multicenter phase II no profit study investigating the disease-free survival efficacy of niraparib as maintenance treatment in 46 patients with metastatic colorectal cancer with partial or complete response after oxaliplatin-based induction therapy.

The study also includes translational research objectives.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years at time of study entry
* Histologically confirmed diagnosis of Stage IV colorectal adenocarcinoma
* Disease evaluation with proven Complete Response or Partial Response according to RECIST v 1.1 after 4 months of oxaliplatin-based doublets or triplets with or without anti-VEGF or anti-EGFR agents
* Availability of Formalin-Fixed Paraffin-Embedded tumor tissue
* Treatment with Niraparib must be started after at least 2 weeks the end of platinum-based induction therapy up to 6 weeks
* Eastern Cooperative Oncology Group Performance Status < 1
* Adequate normal organ and marrow function as follow: Haemoglobin≥9.0 g/dL; b. Absolute neutrophil count ≥1.5 × 109 /L; Platelet count ≥100 × 109/L; Serum bilirubin ≤1.5 x Upper Limit of Normal This will not apply to patients with Gilbert's syndrome; Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula; Aspartate aminotransferase /Alanine Aminotransferase ≤2.5 x Upper Limit of Normal o ≤ 5 x Upper Limit of Normal in the presence of liver metastases
* Willing and able to comply with all of the requirements and visits in the protocol
* Participant must agree not to donate blood during the study or for 90 days after the last dose of Niraparib
* Fertile women must have a negative urine or serum pregnancy test within 7 days prior to taking study treatment
* Fertile women must use highly effective contraception, starting with the screening visit through 6 months post last dose of Niraparib.
* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 90 days after the last dose of study treatment.
* Male participant must not donate sperm for 90 days after last dose of Niraparib.

Exclusion Criteria:

* Prior adjuvant treatment for stage II/III colorectal cancer ending within 12 months before the start of induction treatment
* Patients with Microsatellite instability high or DNA mismatch repair deficiency DSBs DNA double-strand breaks are not allowed
* Any systemic disease that, in the opinion of the Investigator, it is not compatible with the protocol
* Major surgery ≤ 3 weeks prior to initiating Niraparib
* Participation in another interventional clinical trial
* Radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy < 1 week prior to taking Niraparib
* Hypersensitivity to Niraparib components or excipients
* Transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating Niraparib
* Colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior Niraparib
* Any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks
* History of myelodysplastic syndrome, acute myeloid leukemia or Prior Reversible Encephalopathy Syndrome
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection.
* Diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating Niraparib (except basal or squamous cell carcinoma of the skin and cervical cancer in situ that has been definitively treated)
* Active infection with Human Hepatitis B Virus or Hepatitis C Virus
* Pregnancy or breastfeeding
* Any impairment of gastrointestinal function or disease that may significantly impair the absorption of oral drugs, malabsorption syndrome, bowel obstruction, or inability to swallow tablets).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival 1 | 36 months
  Progression-Free Survival 1 is defined as the time from the patient registration to the date of first radiographic progression by RECIST guidelines (version 1.1), or death from any cause in the absence of progression, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival (2) after re-introduction of first-line treatment combination | 36 months
  Progression-Free Survival (2) is defined as the patient registration to progression or death from any cause in the absence of progression, whichever comes first on anticancer treatment following maintenance therapy.
Overall Survival | 36 months
  Overall Survival is defined as time from patient registration until death from any cause. If no event (death) has been observed, the patient is censored at the date of last follow up
Objective Response Rate | 36 months
  Objective Response Rate is defined as the percentage of patients with Complete Response or Partial Response, as assessed by Response Evaluation Criteria in Solid Tumors v.1.1 criteria using an independent review.
Incidence of Treatment-Emergent Adverse Events | 36 months
  Toxicity / adverse events classified according to NCI-Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Translational objectives for evaluated Association between DNA damage responseprotein expression with Progression-free survival of Niraparib maintenance | 36 months
  Association between DNA damage responseprotein expression with Progression-free survival of Niraparib maintenance
Translational objectives 2 for evaluated association of Colorectal Cancer-optimized mutational signatures, including HRDetect, with Progression-free survival of Niraparib maintenance | 36 months
  Association of Colorectal Cancer-optimized mutational signatures, including HRDetect, with Progression-free survival of Niraparib maintenance
Translational objectives 3 for evaluated association between in vitro drug screening sensitivity on Patient-derived organoids and clinical outcome | 36 months
  Association between in vitro drug screening sensitivity on Patient-derived organoids and clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sobrero, Principal Investigator — Ospedale Policlinico San Martino IRCCS; Alberto Puccini, Study Chair — Ospedale Policlinico San Martino IRCCS